CLINICAL TRIAL: NCT01072630
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dosage Study to Evaluate the Efficacy and Safety of Armodafinil Treatment (150 and 200 mg/Day) as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Brief Title: Study to Evaluate the Efficacy and Safety of Armodafinil Treatment as Adjunctive Therapy in Adults With Major Depression Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C10953/3072; 2009-016634-27 (EudraCT Number)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Depression
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Depression | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants were administered placebo and titrated to match the armodafinil treatment arms. Total treatment was 8 weeks.
  Interventions: Drug: Placebo
- Armodafinil 150 mg/day (Experimental): Participants started the study at a dose of 50mg/day of armodafinil and titrated up in the first week to 150 mg/day. The 150 mg/day dosage was continued for 7 more weeks for a total of 8 weeks of treatment.
  Interventions: Drug: Armodafinil
- Armodafinil 200 mg/day (Experimental): Participants started the study at a dose of 50mg/day of armodafinil and titrated up in the first week to 200 mg/day. The 200 mg/day dosage was continued for 7 more weeks for a total of 8 weeks of treatment. This treatment arm was discontinued via a protocol amendment.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — Doses of either 150mg/day or 200 mg/day in tablet form taken orally, once daily in the morning.
  Other Names: Nuvigil; CEP-10953
  Arms: Armodafinil 150 mg/day; Armodafinil 200 mg/day
Drug: Placebo — Matching Placebo, also in tablet form taken orally, once daily in the morning.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine whether armodafinil treatment, at a dosage of 150 mg/day, is more effective than placebo treatment as adjunctive therapy to mood stabilizers for treatment of adults with major depression associated with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of bipolar I disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria and is currently experiencing a major depressive episode.
* Documentation that the patient has had at least 1 previous manic or mixed episode.
* The patient has had no more than 6 mood episodes in the last year.
* The patient's current major depressive episode must have started no less than 2 weeks and no more than 12 months prior to the screening visit. The current depressive episode must have begun after the patient's current mood stabilizer regime began.
* The patient must have been taking 1 (or 2) of the following protocol-allowed mood stabilizers: lithium, valproic acid, lamotrigine, aripiprazole, olanzapine, risperidone, or ziprasidone (only if taken in combination with lithium or valproic acid).
* Written informed consent is obtained.
* The patient is a man or woman 18 through 65 years of age.
* The patient is in good health (except for diagnosis of bipolar I disorder) as judged by the investigator, on the basis of medical and psychiatric history, medical examination, electrocardiography (ECG), serum chemistry, hematology, and urinalysis.
* Women of childbearing potential (women who have not reached menopause, women who are less than 2 years postmenopausal, and women who are not surgically sterile) who are sexually active must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study.
* The patient is willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.
* The patient has permanent accommodations and means of being contacted by the study center.
* The patient understands that they may enroll in this clinical study only once and may not enroll in any other clinical study while participating in this trial.

Exclusion Criteria:

* The patient has any Axis I disorder apart from bipolar I disorder that was the primary focus of treatment within 6 months of the screening visit or during the screening period.
* The patient has psychotic symptoms or has had psychosis within 4 weeks of the screening visit or during the screening period.
* The patient has current active suicidal ideation, is at imminent risk of self-harm, or has a history of significant suicidal ideation or suicide attempt at any time in the past that causes concern at present.
* The patient has a history of an eating disorder or obsessive compulsive disorder (OCD) within 6 months of the screening visit or during the screening period.
* The patient has a history of alcohol or substance abuse or dependence (with the exception of nicotine dependence) within 3 months of the screening visit or during the screening period.
* The patient has a history of any cutaneous drug reaction or drug hypersensitivity reaction, a history of any clinically significant hypersensitivity reaction, or a history of multiple clinically relevant allergies.
* The patient has any clinically significant uncontrolled medical condition, treated or untreated.
* The patient has received modafinil or armodafinil within the past 5 years, or the patient has a known sensitivity to any ingredients in the study drug tablets.
* The patient has previously participated in a clinical study with armodafinil or has used any investigational product within 90 days of screening. The patient may not enroll in any other clinical study while participating in this study.
* The patient has ever been treated with vagus nerve stimulation (VNS) or deep brain stimulation (DBS), or has been treated with electroconvulsive therapy (ECT) or repetitive transcranial magnetic stimulation (rTMS) within 3 months of the screening visit.
* The patient is a pregnant or lactating woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (92):
- United States (46):
  - Birmingham Psychiatry Pharmaceutical Studies, Inc, Birmingham, Alabama
  - South Coast Medical Associates/SC Clinical Trials, Inc., Anaheim, California
  - Comprehensive NeuroScience, Cerritos, California
  - Sun Valley Behavioral Medical, Imperial, California
  - North County Clinical Research, Oceanside, California
  - CNRI Los Angeles LLC, Pico Rivera, California
  - CNRI-San Diego LLC, San Diego, California
  - Clinical Innovations Inc., Santa Ana, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Stanford University Medical Center, Stanford, California
  - Viking Clinical Research Center, Temecula, California
  - Comprehensive NeuroScience, Washington D.C., District of Columbia
  - Scientific Clinical Research, Inc., Aventura, Florida
  - Florida Clinical Research Center, Bradenton, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Fidelity Clinical Research, Lauderhill, Florida
  - Compass Research, LLC, Orlando, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Carman Research, Smyrna, Georgia
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Midwest Center for Neurobehavioral Medicine, Oakbrook Terrace, Illinois
  - CNS - Comprehensive Neuro Science, Park Ridge, Illinois
  - Community Research, Crestview Hills, Kentucky
  - AccelRx Research, Fall River, Massachusetts
  - Mayo College of Medicine, Rochester, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - CRI Worldwide, LLC, Mount Laurel, New Jersey
  - Behavioral Medical Research of Brooklyn, Brooklyn, New York
  - Fieve Clinical Services, Inc., New York, New York
  - Medical and Behavioral Health Research, New York, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - North Coast Clinical Trials, Inc., Beachwood, Ohio
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigators, Inc. (OCCI, Inc.), Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Belmont Center for Comprehensive Treatment, Philadelphia, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Insite Clinical Research, DeSoto, Texas
  - Red Oak Psychiatry Associates, P.A., Houston, Texas
  - University Hills Clinical Research, Irving, Texas
  - Aspen Clinical Research, LLC, Orem, Utah
  - Clinical Methods, Salt Lake City, Utah
  - Alliance Research Group, Richmond, Virginia
- Argentina (6):
  - Dr. Gregorio Hugo Sorin, Buenos Aires, Buenos Aires
  - INECO, Buenos Aires, Buenos Aires
  - Instituto FLENI, Buenos Aires, Buenos Aires
  - Sanatorio Prof. León S. Morra SA, Córdoba, Córdoba Province
  - Centro de Investigación y asistencia en Psiquiatria (CIAP), Rosario, Rosario
  - B.A. Psychiatric Research Cent, Buenos Aires
- Australia (2):
  - Neurotherapy Victoria Clinical Trials, Malvern, Victoria
  - Northern Area Mental Health Services Northern Psychiatric R, Melbourne, Victoria
- Bulgaria (8):
  - MHAT Doverie, Sofia, Sofia
  - Psychiatric clinic, University Hospital "Alexandrovska", Sofia, Sofia
  - MHAT - Sveta Marina, Varna, Varna
  - District Department of Psychiatric Disorders With Stationary, Burgas
  - State Psychiatric Hospital - Pazardjik, Pazardzhik
  - Psychiatric clinic for women UMHAT "Dr. Georgi Stranski", Pleven
  - ODPZS- EOOD, Plovdiv, Bulgaria, Plovdiv
  - Diagnostic Consultative Center "Tchaika", Varna
- Canada (5):
  - Grey Nuns Hospital, Edmonton, Alberta
  - Dr. Alexander McIntyre, Inc., Penticton, British Columbia
  - Providence Care Mental Health Services, Kingston, Ontario
  - Medical Research Associates, Mississauga, Ontario
  - Hôpital Louis Hlafontaine, Montreal, Quebec
- France (3):
  - CMP/CHS du Jura, Dole
  - Centre Hospitalier de Jonzac, Jonzac
  - Hopital Universitaire Caremeau-Batiment Polyvalent, Service, Nîmes
- Poland (4):
  - Szpital Uniwersytecki im.dr.A.Jurasza w Bydgoszczy, Bydgoszcz, Bydgoszcz
  - Klinika Chorob Psychicznych i Zaburzen Nerwicowych GUM, Gdansk
  - Wojewodzki Szpital Psychiatryczny im. prof. Tadeusza Bilikie, Gdansk
  - Malopolskie Centrum Medyczne, Krakow
- South Africa (7):
  - Cape Trial Centre, Cape Town
  - Flexivest Fourteen Research Centre, Cape Town
  - Knighton Surgery, Cape Town
  - Vista Clinic, Centurion
  - Dr Magnus & Dr Brink, Johannesburg
  - Paarl Medical Centre, Paarl
  - Dey Clinic, Pretoria
- Spain (4):
  - Hospital del Henares, Coslada (Madrid)
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital Psiquiátrico de Álava, Vitoria-Gasteiz
  - Hospital Santiago Apostol, Vitoria-Gasteiz
- Ukraine (7):
  - Danylo Galitsky Lviv State Medical University, Lviv, Lviv Oblast
  - Odessa Regional Mental Hospital #2, S. Oleksandrivka, Odesa Oblast
  - Vinnytsa National Medical University named by M.I. Pirogov, Vinnitsa, Vinnitsa
  - Donetsk National Medical University n.a. M. Horkyy, Donetsk
  - Public Institution "Institute of Neurology, Psychiatry and N, Kharkiv
  - Kiev City Psychoneurological Hospital N 1, CNTRP, Kiev
  - Odessa Regional Psychoneurology Dispensary, Odesa

REFERENCES:
- [Derived] Ketter TA, Yang R, Frye MA. Adjunctive armodafinil for major depressive episodes associated with bipolar I disorder. J Affect Disord. 2015 Aug 1;181:87-91. doi: 10.1016/j.jad.2015.04.012. Epub 2015 Apr 15. PMID 25933099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Region 1: USA and Canada Region 2: Eastern European countries, Kyrgyzstan, Mongolia, Uzbekistan, Cyprus, Greece, and Turkey Region 3: Central and Northern European countries, Andorra, Australia, Iceland, Malta, Monaco, San Marino, and Vatican City Region 4: Rest of World
Pre-assignment Details: Participants were randomized (1:1) to receive150 mg/day armodafinil or matching placebo. The 200-mg/day armodafinil treatment group was discontinued per protocol Amendment 03. Randomization was stratified on the basis of the mood-stabilizing medication and region of the world.
Period: Overall Study
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Started | 230 | 232 | 30
Safety Population | 229 (Treated participants. One participant was randomized but not treated.) | 231 (Treated participants. One participant was randomized but not treated.) | 30 (Treated participants.)
Full Analysis Population | 224 (Treated participants who have at least 1 postbaseline IDS-C30 efficacy assessment) | 230 (Treated participants who have at least 1 postbaseline IDS-C30 efficacy assessment) | 28 (Treated participants who have at least 1 postbaseline IDS-C30 efficacy assessment)
Completed | 175 | 172 | 17
Not Completed | 55 | 60 | 13
Not completed — Adverse Event | 11 | 19 | 2
Not completed — Lack of Efficacy | 10 | 10 | 1
Not completed — Withdrawal by Subject | 8 | 7 | 2
Not completed — Protocol Violation | 10 | 8 | 4
Not completed — Lost to Follow-up | 11 | 11 | 1
Not completed — Noncompliance with study medication | 1 | 1 | 1
Not completed — Noncompliance with study procedures | 1 | 2 | 1
Not completed — Other | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day | Total
Number analyzed (Participants) | 230 | 232 | 30 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.52) | 44.4 (11.00) | 41.2 (12.60) | 43.9 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 128 | 20 | 273
  Male | 105 | 104 | 10 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 2 | 36
  Not Hispanic or Latino | 203 | 206 | 28 | 437
  Unknown or Not Reported | 9 | 10 | 0 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 54 | 49 | 13 | 116
  White | 162 | 166 | 14 | 342
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 15 | 1 | 25
Weight [Mean (Standard Deviation); unit: kg] | 86.7 (20.21) | 86.3 (19.21) | 96.7 (21.91) | 87.1 (19.96)
Height [Mean (Standard Deviation); unit: cm] | 169.6 (9.88) | 169.9 (9.44) | 170.4 (8.25) | 169.7 (9.57)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.86) | 29.9 (6.39) | 33.6 (7.58) | 30.3 (6.73)
Time Since Start of Current Depressive Episode [Mean (Standard Deviation); unit: weeks] | 11.2 (7.79) | 12.4 (8.99) | 14.7 (8.73) | 12.0 (8.46)
Time Since First Diagnosis for Bipolar [Mean (Standard Deviation); unit: years] | 11.4 (9.57) | 11.7 (9.49) | 13.3 (10.96) | 11.6 (9.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Total Score From the 30-Item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Time Frame: Day 0 (baseline), Week 8
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- All Armodafinil: This arm combines participants who took 150 mg/day and those in the discontinued treatment arm who took 200 mg/day of armodafinil for 8 weeks.
Arm/Group | Placebo | Armodafinil 150 mg/Day | All Armodafinil
Number analyzed (Participants) | 224 | 230 | 258
units on a scale | -18.8 (1.02) | -20.9 (1.02) | -20.7 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Armodafinil 150 mg/Day; Test type: Superiority or Other; p = 0.1302, mixed-model repeated measures (MMRM) — All statistical tests were 2-tailed at the 0.05 level of significance; Treatment, visit, treatment-by-visit interaction, concurrent mood-stabilizing medication, and region of the world used as fixed factors; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-4.67 to 0.60]
Statistical Analysis 2: Comparison: Placebo vs All Armodafinil; Test type: Superiority or Other; p = 0.1350, mixed-model repeated measures (MMRM) — All statistical tests were 2-tailed at the 0.05 level of significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.51 to 0.61]

2. Secondary Outcome: Percentage of Responders At Different Treatment Weeks According to the 30-Item Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) Total Score
Description: A responder is a participant with a ≥50% decrease or greater from baseline in the total score of the IDS-C30. The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. The denominator for calculating the percentages at each visit is the number of participants with a nonmissing value at that visit. Endpoint was the last observed postbaseline data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 224 | 230 | 28
percentage of participants
  Week 1 (218, 223, 27) | 5 | 7 | 22
  Week 2 (209, 212, 25) | 16 | 17 | 20
  Week 4 (193, 190, 22) | 28 | 27 | 41
  Week 6 (182, 181, 18) | 36 | 41 | 56
  Week 7 (172, 178, 14) | 40 | 44 | 57
  Week 8 (172, 169, 17) | 47 | 49 | 59
  Endpoint (224, 230, 28) | 39 | 40 | 39

3. Secondary Outcome: Percentage of Participants in Remission At Different Treatment Weeks According to the 30-Item Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) Total Score
Description: A participant in remission was defined as a participant with an IDS-C30 total score of 11 or less.
  The IDS-C30 is a standardized 30-item, clinician-rated scale to assess the severity of a participant's depressive symptoms. Every effort was made to have the same rater evaluate a participant across all visits.
  Total scores range from 0-84, with a score of 0 indicating no depression and a score of 84 indicating the most severe depression.
Time Frame: Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 224 | 230 | 28
percentage of participants
  Week 1 (218, 223, 27) | .5 | 1 | 7
  Week 2 (209, 212, 25) | 7 | 4 | 12
  Week 4 (193, 190, 22) | 11 | 8 | 18
  Week 6 (182, 181, 18) | 19 | 15 | 39
  Week 7 (172, 178, 14) | 19 | 17 | 43
  Week 8 (172, 169, 17) | 22 | 23 | 47
  Endpoint (224, 230, 28) | 17 | 18 | 29

4. Secondary Outcome: Change From Baseline to Different Treatment Weeks in the Total Score From the 30-Item Inventory of Depressive Symptomatology-Clinician-Rated (IDS-C30)
Description: as for outcome 1
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. Participants are included in the analysis at each timepoint if they have a nonmissing value at that visit. Endpoint for analyses was the last observed postbaseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 224 | 230 | 28
units on a scale
  Week 1 (218, 223, 27) | -6.6 (7.59) | -7.2 (8.28) | -9.9 (12.92)
  Week 2 (209, 212, 25) | -11.1 (10.72) | -11.8 (9.85) | -13.9 (11.99)
  Week 4 (193, 190, 22) | -15.1 (12.14) | -16.7 (10.98) | -17.8 (12.82)
  Week 6 (182, 181, 18) | -18.1 (12.60) | -19.1 (11.77) | -20.7 (12.30)
  Week 7 (172, 178, 14) | -19.0 (13.38) | 021.0 (12.12) | -22.8 (14.57)
  Week 8 (172, 169, 17) | -20.2 (13.81) | -22.4 (12.63) | -21.8 (13.42)
  Endpoint (224, 230, 28) | -17.5 (14.28) | -19.1 (13.55) | -18.6 (13.76)

5. Secondary Outcome: Change From Baseline to Different Treatment Weeks in the Total Score From the 16-Item Quick Inventory of Depressive Symptomatology-Clinician-Rated (QIDS-C16)
Description: The QIDS-C16 was derived from specified items in the IDS-C30, clinician-rated scale to assess the severity of a participant's depressive symptoms. Total scores range from 0-27, with a score of 0 indicating no depression and a score of 27 indicating the most severe depression. Negative change from baseline values indicate improvement in the severity of depression.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. The number of participants at each visit is those with a nonmissing value at that visit. Endpoint was the last observed postbaseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 224 | 230 | 28
units on a scale
  Week 1 (218, 223, 27) | -2.7 (3.05) | -2.9 (3.51) | -4.5 (5.16)
  Week 2 (209, 212, 25) | -4.2 (4.02) | -4.5 (3.97) | -6.0 (4.63)
  Week 4 (193, 190, 22) | -5.7 (4.68) | -6.5 (4.29) | -7.4 (4.80)
  Week 6 (182, 181, 18) | -6.8 (4.87) | -7.5 (4.58) | -8.8 (5.05)
  Week 7 (172, 178, 14) | -7.2 (5.13) | -8.1 (4.68) | -9.6 (5.50)
  Week 8 (172, 169, 17) | -7.7 (5.42) | -8.6 (4.88) | -9.8 (5.68)
  Endpoint (224, 230, 28) | -6.7 (5.51) | -7.4 (5.24) | -8.1 (5.47)

6. Secondary Outcome: Change From Baseline to Different Treatment Weeks in the Clinical Global Impression of Severity (CGI-S) for Depression
Description: The CGI-S is an observer-rated scale that measures illness severity on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). Negative change from baseline values indicate improvement in the severity of depression.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: Full analysis set which includes participants who took 1 or more doses of study drug and who have at least 1 postbaseline IDS-C30 efficacy assessment. The number of participants is those with a nonmissing value at that visit. Endpoint was the last observed postbaseline data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 224 | 230 | 28
units on a scale
  Week 1 (218, 223, 27) | -0.2 (0.48) | -0.3 (0.58) | -0.6 (0.97)
  Week 2 (209, 212, 25) | -0.6 (0.83) | -0.6 (0.74) | -0.8 (1.00)
  Week 4 (193, 190, 22) | -0.9 (0.99) | -0.9 (0.90) | -1.1 (1.02)
  Week 6 (182, 181, 18) | -1.1 (1.14) | -1.1 (1.04) | -1.3 (0.97)
  Week 7 (172, 178, 14) | -1.3 (1.14) | -1.3 (1.08) | -1.4 (1.22)
  Week 8 (174, 171, 17) | -1.4 (1.24) | -1.5 (1.13) | -1.8 (1.15)
  Endpoint (224, 230, 28) | -1.2 (1.27) | -1.2 (1.19) | -1.3 (1.21)

7. Secondary Outcome: Change From Baseline to Weeks 4, 8 and Endpoint in the Global Assessment for Functioning (GAF) Scale
Description: The Global Assessment of Functioning (GAF) is a numeric scale (1 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults, e.g., how well or adaptively one is meeting various problems-in-living. Ratings of 1 - 10 mean the participant is in persistent danger of severely hurting self or others (e.g., recurrent violence) or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death. Ratings of 91 - 100 indicate no symptoms, and the participant exhibits superior functioning in a wide range of activities, life's problems never seem to get out of hand, is sought out by others because of his or her many positive qualities. Positive change from baseline values indicate improvement in functioning.
Time Frame: Day 0 (baseline), Weeks 1, 2, 4, 6, 7, and 8, and last postbaseline observation (up to 8 weeks)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 224 | 230 | 28
units on a scale
  Week 4 (193, 190, 22) | 6.4 (8.74) | 7.2 (10.63) | 10.0 (9.74)
  Week 8 (172, 171, 17) | 10.8 (11.01) | 11.6 (11.22) | 13.4 (11.14)
  Endpoint (213, 219, 25) | 9.6 (11.44) | 9.3 (11.85) | 10.5 (10.60)

8. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: AEs were graded by the investigator for severity on a three-point scale: mild, moderate and severe. Causality is graded as either related or not related. A serious adverse event (SAE) is an AE resulting in death, a life-threatening adverse event, hospitalization, a persistent or significant disability/incapacity, a congenital anomaly/birth defect, or an important medical event that may require medical intervention to prevent any of the previous results.
  Protocol-defined adverse events requiring expedited reporting included skin rash, hypersensitivity reaction, emergent suicidal ideation or suicide attempt, and psychosis.
Time Frame: Day 1 to Week 9
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 299 | 123 | 21
participants
  >=1 adverse event | 102 | 123 | 21
  Severe adverse event | 7 | 7 | 1
  Treatment-related adverse event | 59 | 78 | 16
  Deaths | 0 | 1 | 0
  Other serious adverse events | 1 | 5 | 2
  Withdrawn from study due to adverse events | 11 | 19 | 2
  Protocol-defined adverse events | 5 | 3 | 3

9. Secondary Outcome: Change From Baseline to Endpoint in the Young Mania Rating Scale Total Score
Description: The YMRS is a clinician-rated, 11-item checklist used to measure the severity of manic episodes. Information for assigning scores is gained from the participant's subjective reported symptoms over the previous 48 hours and from clinical observation during the interview. Seven items are ranked 0 through 4 and have descriptors associated with each severity level. Four items (irritability, speech, content, and disruptive-aggressive behavior) are scored 0 through 8 and have descriptors for every second increment. The total scale is 0-60. A score of ≤12 indicates remission of manic symptoms, and higher scores indicate greater severity of mania. Negative change from baseline scores indicate a decrease in severity of mania.
Time Frame: Day 0 (baseline), Week 8 or last postbaseline observation (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 226 | 230 | 28
units on a scale | -0.6 (2.76) | -0.5 (3.47) | -0.5 (2.71)

10. Secondary Outcome: Change From Baseline to Endpoint in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: HAM-A measures the severity of anxiety symptoms. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Negative change from baseline scores indicate a decrease in severity of anxiety.
Time Frame: Day 0 (baseline), Week 8 or last postbaseline observation (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. The number analyzed includes participants with both baseline and during treatment assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 218 | 221 | 25
units on a scale | -4.3 (4.95) | -4.0 (5.50) | -2.6 (5.67)

11. Secondary Outcome: Change From Baseline to Endpoint in the Insomnia Severity Index (ISI) Total Score
Description: The ISI is a participant-rated, 7-item questionnaire designed to assess the severity of the participant's insomnia. Each item is ranked 0 (none) through 4 (very severe) and has a descriptor associated with each severity level. Total range is 0 (no insomnia) to 28 (very severe insomnia). Responses to each item are added to obtain a total score to determine the severity of insomnia. Negative change from baseline scores indicate a decrease in severity of insomnia.
Time Frame: Day 0 (baseline), Week 8 or last postbaseline observation (up to 8 weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 217 | 219 | 25
units on a scale | -5.2 (6.89) | -6.7 (7.18) | -6.2 (6.93)

12. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Actual Attempt Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation. The Suicidal Behavior - Actual Attempt question records whether the participant committed a potentially self-injurious act with at least some wish to die since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. The number analyzed includes participants with treatment assessments at the indicated time period.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 0 | 0 | 0

13. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Non-Suicidal Self-Injurious Behavior Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Non-Suicidal Self-Injurious Behavior question records whether the participant committed a potentially self-injurious act that was not associated with a wish to die since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 0 | 0 | 0

14. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Interrupted Attempt Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Interrupted Attempt question records whether the participant was interrupted by an outside circumstance from starting the potentially self-injurious act with at least some wish to die since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 1 | 0 | 0

15. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Aborted Attempt Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Aborted Attempt question records whether the participant began to take steps toward making a suicide attempt but stops themselves before starting the potentially self-injurious act since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 0 | 0 | 0

16. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Suicidal Behavior Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Suicidal Behavior question records whether in the clinician's opinion, the participant exhibited suicidal behavior since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 0 | 0 | 0

17. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Preparatory Acts or Behavior Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Preparatory Acts or Behavior question records whether the participant exhibited acts or preparations towards imminently making a suicide attempt since the last visit.
  .
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 0 | 0 | 0

18. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Behavior - Completed Suicide Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Behavior - Completed Suicide question records whether the participant intentionally causing his/her's own death since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 0 | 0
  Week 2 (209, 212, 25) | 0 | 0 | 0
  Week 4 (193, 190, 22) | 0 | 0 | 0
  Week 6 (182, 181, 18) | 0 | 0 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 0 | 0
  Endpoint (226, 230, 28) | 0 | 0 | 0

19. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Wish to Be Dead Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Wish to Be Dead question records whether the participant endorses thoughts about a wish to dead or not alive anymore, or a wish to fall asleep and not wake up since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 10 | 11 | 2
  Week 2 (209, 212, 25) | 7 | 11 | 0
  Week 4 (193, 190, 22) | 4 | 9 | 0
  Week 6 (182, 181, 18) | 6 | 6 | 0
  Week 7 (172, 178, 14) | 3 | 3 | 0
  Week 8 (174, 171, 17) | 3 | 5 | 1
  Endpoint (226, 230, 28) | 7 | 10 | 2

20. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Non-Specific Active Suicidal Thoughts Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Non-Specific Active Suicidal Thoughts question records whether the participant shares general non-specific thoughts of wanting to end one's life/commit suicide since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (218, 223, 27) | 0 | 2 | 1
  Week 2 (209, 212, 25) | 0 | 1 | 0
  Week 4 (193, 190, 22) | 1 | 1 | 0
  Week 6 (182, 181, 18) | 0 | 3 | 0
  Week 7 (172, 178, 14) | 0 | 0 | 0
  Week 8 (174, 171, 17) | 0 | 1 | 0
  Endpoint (226, 230, 28) | 2 | 2 | 1

21. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Any Methods (Not Plan) Without Intent to Act Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Any Methods (Not Plan) Without Intent to Act question records whether the participant endorses thoughts of suicide and has thought of at least one method but has no specific plan of action since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: The safety analysis set includes randomized participants who took 1 or more doses of study drug. This question is asked if the answer to the 'Non-Specific Active Suicidal Thoughts' question was YES, or based on the judgment of the assessor. The number analyzed includes participants with treatment assessments at the indicated time period.
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (9, 10, 1) | 0 | 0 | 0
  Week 2 (6, 10, 0) | 0 | 1 | 0
  Week 4 (4, 8, 0) | 0 | 1 | 0
  Week 6 (5, 7, 0) | 0 | 2 | 0
  Week 7 (3, 3, 0) | 0 | 0 | 0
  Week 8 (2, 5, 0) | 0 | 0 | 0
  Endpoint (18, 21, 1) | 1 | 2 | 0

22. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Some Intent to Act Without a Specific Plan Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Some Intent to Act Without a Specific Plan question records whether the participant has active suicidal thoughts of killing oneself and reports having some intent to act on such thoughts since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (9, 10, 1) | 0 | 0 | 0
  Week 2 (6, 10, 0) | 0 | 0 | 0
  Week 4 (4, 8, 0) | 0 | 0 | 0
  Week 6 (5, 7, 0) | 0 | 0 | 0
  Week 7 (3, 3, 0) | 0 | 0 | 0
  Week 8 (2, 5, 0) | 0 | 0 | 0
  Endpoint (18, 21, 1) | 1 | 0 | 0

23. Secondary Outcome: Columbia-Suicide Severity Rating Scale 'Since Last Visit' Version (C-SSRS-SLV) For Weeks 1, 2, 4, 6, 7, 8, and Endpoint For the Suicidal Ideation - Specific Plan and Intent Question
Description: The C-SSRS is a clinician-rated scale that assesses suicidality from ideation to behaviors and monitors the potential emergence of suicidality in clinical studies. The C-SSRS-B (baseline) was performed at screening and the C-SSRS-SLV ('Since Last Visit') was performed at baseline and weeks 1, 2, 4, 6, 7, and 8 or last postbaseline observation.
  The Suicidal Ideation - Specific Plan and Intent question records whether the participant has active suicidal thoughts of killing oneself with details of plan fully or partially worked out and the participant has some intent to carry out the plan since the last visit.
Time Frame: Weeks 1, 2, 4, 6, 7, 8, and Endpoint (up to 8 weeks)
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Placebo | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day
Number analyzed (Participants) | 229 | 231 | 30
participants
  Week 1 (9, 10, 1) | 0 | 0 | 0
  Week 2 (6, 10, 0) | 0 | 0 | 0
  Week 4 (4, 8, 0) | 0 | 0 | 0
  Week 6 (5, 7, 0) | 0 | 0 | 0
  Week 7 (3, 3, 0) | 0 | 0 | 0
  Week 8 (2, 5, 0) | 0 | 0 | 0
  Endpoint (18, 21, 1) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 9
Arm/Group | Armodafinil 150 mg/Day | Armodafinil 200 mg/Day | Placebo
Serious Adverse Events (participants affected / at risk) | 5/231 | 2/30 | 1/229
Other Adverse Events (participants affected / at risk) | 80/231 | 18/30 | 59/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150 mg/Day (N=231) | Armodafinil 200 mg/Day (N=30) | Placebo (N=229)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil 150 mg/Day (N=231) | Armodafinil 200 mg/Day (N=30) | Placebo (N=229)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 5 (8) | 13 (16)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 5 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (18) | 4 (5) | 5 (5)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 7 (9) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 38 (45) | 4 (5) | 30 (39)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2) | 6 (6)
Insomnia (Psychiatric disorders) | 12 (12) | 4 (5) | 8 (8)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.